CLINICAL TRIAL: NCT01867398
Title: The Investigation of the Impact of Atypical Antipsychotics on Brain Functioning in Youths With Conduct Disorder
Brief Title: Effects of Atypical Antipsychotics on Brain Function in Children and Teens With Conduct Disorders
Status: Terminated | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Collaborators: Boys Town Research Hospital (Unknown)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999913125; 13-M-N125
Record Dates: First submitted 2013-05-31; First posted 2013-06-04 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2015-05-18

CONDITIONS: Conduct Disorder; fMRI
Keywords: Conduct Disorder; Antipsychotic; Treatment Study; Functional Magnetic Resonance Imaging (fMRI); Adolescents
MeSH Terms: conditions — Conduct Disorder

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Some children and teenagers have conditions known as conduct disorders. They often have long-term chronic behavior problems, such as defiant behavior or violence. Conduct disorders are often treated with antipsychotic medication. Researchers want to study two types of newer antipsychotics (aripiprizole and risperidone) for children and adolescents with conduct disorders. They will look at how these drugs affect brain activity. To do so, they will give brain activity tests using magnetic resonance imaging (MRI). The tests will compare the results from healthy volunteer children and teens to those of others with behavior problems.

Objectives:

- To see how atypical antipsychotics affect brain activity of children and teenagers with conduct disorders.

Eligibility:

* Children and teenagers between 10 and 18 years of age who have a conduct disorder and are taking aripiprizole.
* Children and teenagers between 10 and 18 years of age who have a conduct disorder and are taking risperidone.
* Children and teenagers between 10 and 18 years of age who have a conduct disorder and are not taking an atypical antipsychotic.
* Healthy volunteers between 10 and 18 years of age.

Design:

* Participants will be screened with a physical exam and medical history. Parents/guardians will be asked questions about their child s feelings, experiences, and behavior. Participants will also answer questions about their feelings and moods.
* This study will involve two visits. Each visit will involve MRI scanning.
* At the first visit, participants will have memory and thinking tests. The tests will involve making decisions or playing games. Some of these tests will use MRI scanning to look at brain activity.
* The second visit will be 3 to 5 months after the first visit. The tests from the first visit will be repeated.

DETAILED DESCRIPTION:
Objective: To determine the impact, as indexed by BOLD response, of the administration of aripiprazole and risperidone during the treatment of Conduct Disorder (CD) on the pathophysiology of CD.

Study Population: Youth with CD receiving aripiprazole at admission to Boys Town Omaha, youth with CD receiving risperidone at admission to Boys Town Omaha, youth with CD not receiving antipsychotics at admission to Boys Town Omaha, typically developing youth.

Design: The study will involve a 4 (Group: CD receiving aripiprazole at admission, CD receiving risperidone at admission, CD not receiving antipsychotics at admission, typically developing youth) x 2 (Time: At admission vs. four months subsequent to admission [when treatment for the antipsychotic groups will have been tapered off]) design. Principle dependent measures will relate to BOLD response indices of the pathophysiology of CD.

Outcome Measures: Principle dependent measures will relate to BOLD response indices of the pathophysiology of CD. In addition, assessments of symptom severity will be collected, as will measurements of cognitive function.

ELIGIBILITY:
* INCLUSION CRITERIA:

Youth with Conduct Disorder (CD)

1. 10-18 years of age.
2. A current diagnosis of CD.
3. Currently taking aripiprazole, risperidone or unmedicated with antipsychotics.

Typically developing (TD) youth

1. 10-18 years of age.
2. No current psychiatric diagnosis.

EXCLUSION CRITERIA:

1. I.Q.< 80.
2. Pregnancy.
3. Ongoing medical illness requiring the following medications:

   * Beta blockers
   * Steroids
   * Receipt of any antipsychotic medication other than aripiprazole or risperidone.
   * Receipt of risperidone for the CD group medicated with aripiprazole.
   * Receipt of aripiprazole for the CD group medicated with risperidone.
   * Receipt of antipsychotics for the un-medicated CD group.
   * Explicit exclusions include active psychosis, Pervasive Developmental
   * Neurologic disorder (including seizures).
   * Any ferromagnetic metallic objects in the body. Metal plates, certain types of dental braces, cardiac pacemakers, etc., that are sensitive to electromagnetic fields contraindicate MRI scans.
   * Claustrophobia

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2013-04-29; Primary Completion 2015-05-18 (Actual); Study Completion 2015-05-18 (Actual)

PRIMARY OUTCOMES:
Principle dependent measures will relate to BOLD response indices of the pathophysiology of CD. | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: James J Blair, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- Boys Town Research Hospital, Omaha, Nebraska, United States

REFERENCES:
- [Background] Allison DB, Casey DE. Antipsychotic-induced weight gain: a review of the literature. J Clin Psychiatry. 2001;62 Suppl 7:22-31. PMID 11346192
- [Background] Aman MG, De Smedt G, Derivan A, Lyons B, Findling RL; Risperidone Disruptive Behavior Study Group. Double-blind, placebo-controlled study of risperidone for the treatment of disruptive behaviors in children with subaverage intelligence. Am J Psychiatry. 2002 Aug;159(8):1337-46. doi: 10.1176/appi.ajp.159.8.1337. PMID 12153826
- [Background] Bortolozzi A, Diaz-Mataix L, Toth M, Celada P, Artigas F. In vivo actions of aripiprazole on serotonergic and dopaminergic systems in rodent brain. Psychopharmacology (Berl). 2007 Apr;191(3):745-58. doi: 10.1007/s00213-007-0698-y. Epub 2007 Jan 30. PMID 17265076